CLINICAL TRIAL: NCT07314671
Title: Effects of a Dynamic Versus an Isometric Copenhagen Adduction Exercise on Muscle Strength and Athletic Performance in Youth Football: A Randomized Controlled Trial
Brief Title: Isometric vs Dynamic Copenhagen Adduction Exercise in Football Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Christos Pippas, Principal investigator, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 60372/01-07-2025
Record Dates: First submitted 2025-11-19; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Groin Injuries
Keywords: Groin, exercise training, Copenhagen Adduction, football
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The participants will be assigned to either a dynamic (DCA) or an isometric (ICA) Copenhagen Adduction exercise group and perform a progressive exercise protocol for 6 weeks during at the club's training facilities.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Copenhagen Adduction (DCA) (Experimental)
  Interventions: Other: Exercise
- Isometric Copenhagen Adduction (ICA) (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both groups (DCA, ICA) will perform 2 weekly sessions, 2 sets per side, 6-12 repetitions

SUMMARY:
Hip adductor strength training is important for groin injuries rehabilitation and prevention. A widely used exercise is the Copenhagen Adduction (CA) exercise. The current study will include young football players (12-16 yrs) individually randomised into two CA groups (isometric, dynamic) training 2 times per week for 6 weeks. Both groups will use 2 sets per side and a range of 6-12 repetitions. Maximal eccentric (EHAD) and isometric (IHAD) hip adduction torque, jump and sprint capacity, delayed onset muscle soreness (DOMS), and perceived exertion will be recorded. A minimum of 42 participants will be required.

DETAILED DESCRIPTION:
Introduction: Groin injuries are one of the most common injuries in sports such as basketball, hockey and handball. They account for 4-19% of all injuries in Association football (soccer), with movements such as shooting or passing, changes of direction, and jumping being the most common injury mechanisms. Previous groin injury and low hip adductor strength have been shown to be risk factors for groin injuries. Exercise has shown a positive effect on adductor muscle strength, groin pain rehabilitation, and prevention. An exercise widely used in adductor strength training and groin pain rehabilitation is the Copenhagen Adduction (CA) exercise. Another exercise used in groin pain rehabilitation and adductor strength training is the adductor squeeze exercise. Although there are investigations comparing the strength effects of the CA with these of other dynamic exercises, and isometric exercises, there is only one study that included the CA using isometric contraction during a progressive training protocol for the hip adductor muscles, and no studies comparing two contraction types of the CA. Although muscle strengthening is an important component in football training, sprint and jump training also plays an important role in athletes' performance. There is only one study which evaluated the effects of the CA and Nordic Hamstring exercise on athletic performance.

Aim: To compare the effects of a dynamic and an isometric CA on adductor muscle strength and athletic performance (sprint, jump) in male football (soccer) players.

Methods: Young football players (12-16 yrs) will be included in the study. They will be individually randomised into two CA groups (isometric, dynamic) and will train 2 times per week for six weeks using 2 sets per side and a range of 6-12 repetitions maintaining the same repetition number and time under tension. The strength and athletic performance testing will be performed by a physiotherapist and an exercise therapist, respectively. They will not participate in the intervention supervision and will be unaware of the group allocation. The physiotherapist and the exercise therapist who will supervise the intervention, as well as the participants, will not be aware of the testing results until the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

Healthy male soccer players between 12 and 16 years old systematically (≥4 times per week) participating in training and games

Exclusion Criteria:

1. musculoskeletal injury and/or neurological disorder that would affect strength and/or athletic performance testing, and/or exercise execution.
2. adductor muscle injury within 6 months before study initiation.
3. groin pain greater than 2/10 on a Numeric Rating Scale (NRS) during strength and/or athletic performance testing, and/or during exercise execution.
4. any systematic strength training of the adductor muscles during the last month prior to study initiation.

Ages: 12 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Eccentric hip adductor torque | From enrollment to the end of treatment at 6 weeks
  Maximal eccentric (EHAD) hip adduction torque. Players' strength will be measured in Newtons, leg length in centimeters, and weight in kilograms. These measures will be combined for eccentric torque (Nm/kg) to be recorded and analysed.
Isometric hip adduction torque | From enrollment to the end of treatment at 6 weeks
  Maximal isometric (IHAD) hip adduction torque. Players' strength will be measured in Newtons, leg length in centimeters, and weight in kilograms. These measures will be combined for isometric torque (Nm/kg) to be recorded and analysed.

SECONDARY OUTCOMES:
Jump performance | From enrollment to the end of treatment at 6 weeks
  Jump (squat jump, countermovement jump, countermovement jump with arm swing) capacity will be measured in centimetres.
Sprint capacity | From enrollment to the end of treatment at 6 weeks
  Sprint (5 meters, 10 meters, 20 meters) capacity will be measured in seconds.
Delayed onset muscle soreness | From enrollment to the end of treatment at 6 weeks
  Delayed onset muscle soreness (DOMS) will be recorded with the use of a numeric rating scale 0-10.
Perceived exertion | From enrollment to the end of treatment at 6 weeks
  Perceived exertion will be recorded with the use of a numeric rating scale 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Pippas, Principal Investigator — University of West Attica

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the corresponding author upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: Beginning after publication with no end date
Access Criteria: The data that support the findings of this study will be available from the corresponding author upon reasonable request
URL: http://datarepository.will-be-provided-after-study-completion

REFERENCES:
- [Background] Polglass G, Burrows A, Willett M. Impact of a modified progressive Copenhagen adduction exercise programme on hip adduction strength and postexercise muscle soreness in professional footballers. BMJ Open Sport Exerc Med. 2019 Oct 15;5(1):e000570. doi: 10.1136/bmjsem-2019-000570. eCollection 2019. PMID 31673404
- [Background] Serner A, Jakobsen MD, Andersen LL, Holmich P, Sundstrup E, Thorborg K. EMG evaluation of hip adduction exercises for soccer players: implications for exercise selection in prevention and treatment of groin injuries. Br J Sports Med. 2014 Jul;48(14):1108-14. doi: 10.1136/bjsports-2012-091746. Epub 2013 Mar 19. PMID 23511698
- [Background] Pippas C, Gioftsos G, Korakakis V, Serner A. Strength effects of the Copenhagen adduction exercise vs an adductor squeeze exercise in male football players - A randomized controlled trial. Sci Med Footb. 2025 Nov;9(4):382-391. doi: 10.1080/24733938.2024.2419659. Epub 2024 Oct 24. PMID 39444266
- [Background] Haroy J, Thorborg K, Serner A, Bjorkheim A, Rolstad LE, Holmich P, Bahr R, Andersen TE. Including the Copenhagen Adduction Exercise in the FIFA 11+ Provides Missing Eccentric Hip Adduction Strength Effect in Male Soccer Players: A Randomized Controlled Trial. Am J Sports Med. 2017 Nov;45(13):3052-3059. doi: 10.1177/0363546517720194. Epub 2017 Aug 14. PMID 28806100
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28806100/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39444266/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31673404/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23511698/
- Available data/document: Protocol background: 10.1136/bjsports-2012-091746 — https://pubmed.ncbi.nlm.nih.gov/23511698/
- Available data/document: Protocol background: 10.1136/bmjsem-2019-000570 — https://pubmed.ncbi.nlm.nih.gov/31673404/
- Available data/document: Protocol background: 10.1080/24733938.2024.2419659 — https://pubmed.ncbi.nlm.nih.gov/39444266/
- Available data/document: Protocol background: 10.1177/0363546517720194 — https://pubmed.ncbi.nlm.nih.gov/28806100/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT07314671/Prot_SAP_000.pdf